CLINICAL TRIAL: NCT05309824
Title: Cognitive Dysfunction in Cardiovascular Patients Based on Resting fMRI
Brief Title: Cardiovascular Disease Cohort
Status: Withdrawn | Type: Observational
Why Stopped: The study was stopped due to the COVID-19 situation.
Sponsor: Westlake University (Other)
Collaborators: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: 20220303ZJS001
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Decline; Cardiovascular Diseases
MeSH Terms: conditions — Cognitive Dysfunction; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool and saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Atrial fibrillation
- Left ventricular hypertrophy
- Pulmonary hypertension
- Coronary atherosclerotic heart disease
- Heart failure with retained ejection fraction

SUMMARY:
The Cardiovascular Disease Cohort study is a prospective cohort study among cardiovascular disease patients enrolled in the Affiliated Hospital of Hangzhou Normal University. The primary aim of this study is to explore the brain mechanism of cognitive decline in cardiovascular disease patients using RS-FMRI and multi-omics techniques (including microbiome and metabolomics). Another aim of this study is to develop diagnosis and treatment strategies combining cardiovascular disease and cognitive function.

ELIGIBILITY:
1. Atrial fibrillation patients

   Inclusion Criteria:
   * Age: 45-80 years old;
   * Consistent with the diagnosis of atrial fibrillation: standard 12-lead ECG recording or ≥30s single-lead ECG recording or 24-hour dynamic electrocardiogram, no obvious repeated P wave, irregular RR interval (when it does not damage atrioventricular conduction) can be diagnosed as clinical atrial fibrillation;
   * Anticoagulant therapy was selected according to cha2DS2-VASC score and HASBLED score;
   * Voluntarily participate in the study and sign the informed consent.

   Exclusion Criteria:
   * Valvular atrial fibrillation, atrial fibrillation caused by hyperthyroidism;
   * Severe liver and kidney failure;
   * Malignant tumor;
   * Diseases of the blood system;
   * History of major surgical trauma within six months.
2. Left ventricular hypertrophy patients

   Inclusion Criteria:
   * Age: 45-80 years old;
   * ECG diagnosis of left ventricular hypertrophy: increased QRS group voltage: CHEST lead Rv5 or Rv6>2.5mV; Rv5+Sv1>4.0mV (male) or >3.5mV (female) Or in the limb lead, R1>11.5 mV; RaVL > 1.2 mV; RaVF > 2.0 mV; RI + SIII > 2.5 mV;
   * Sign informed consent to participate in the study voluntarily.

   Exclusion Criteria:
   * Left ventricular hypertrophy caused by valvular heart disease and hyperthyroidism;
   * Severe liver and kidney failure;
   * Malignant tumor;
   * Diseases of the blood system;
   * History of major surgical trauma within six months.
3. Pulmonary hypertension patients

   Inclusion Criteria:
   * Age: 18-80 years;
   * Consistent with the diagnosis of pulmonary hypertension: at sea level and resting state, average pulmonary arterial pressure (mPAP) ≥25 mmHg (1mmHg=0.133kPa) measured by right heart catheter, or pulmonary arterial pressure ≥35 mmHg estimated by tricuspid regurgitation velocity indicated by cardiac ultrasound;
   * Sign informed consent to participate in the study voluntarily.

   Exclusion Criteria:
   * Patients with other serious cardiovascular and cerebrovascular diseases;
   * Severe liver and kidney failure;
   * Malignant tumor;
   * Diseases of the blood system;
   * History of major surgical trauma within six months.
4. Patients with coronary atherosclerotic heart disease

   Inclusion Criteria:
   * Age: 45-80 years old;
   * In line with the diagnosis of coronary heart disease: coronary artery stenosis indicated by CORONARY CTA or angiography, with a severity of more than 50%, accompanied by symptoms of chest distress and chest pain;
   * Sign informed consent to participate in the study voluntarily.

   Exclusion Criteria:
   * Severe valvular heart disease, hyperthyroidism, etc;
   * Severe liver and kidney failure;
   * Malignant tumor;
   * Diseases of the blood system;
   * History of major surgical trauma within six months.
5. Heart failure with retained ejection fraction patients

Inclusion Criteria:

* Age: 45-80 years;
* Patients with HFpEF diagnosis had clinical symptoms or signs of cardiac insufficiency, cardiac echocardiography suggested left ventricular eject fraction (LVEF≥50%), increased natriuretic peptide, and met at least one of the following criteria: a. Left ventricular hypertrophy and/or left atrium enlargement; B. Abnormal diastolic function of the heart.
* It is necessary to rule out that the patient's symptoms are not caused by heart disease; ④ Voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

* Severe cervical and cerebrovascular events, such as severe carotid artery plaque or stenosis (stenosis rate greater than 50%), cerebral ischemic stroke, etc;
* Severe liver and kidney failure;
* Malignant tumor;
* Diseases of the blood system;
* History of major surgical trauma within six months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with five types of cardiovascular diseases (atrial fibrillation, left ventricular hypertrophy, pulmonary hypertension, coronary heart disease, and heart failure with retained ejection fraction) are planned to be enrolled in the Affiliated Hospital of Hangzhou Normal University.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
MMSE | Baseline
  The investigators assessed orientation (10 points), immediate recall (3 points), attention and computation (5 points), delayed recall (3 points), language function (8 points) (naming, retelling, reading, writing, understanding), and visuospatial perception (1 point). The total score is 30 points, and the demarcation between normal and abnormal is related to education level: the uneducated ≤17 points, the primary school group ≤6 years of education ≤20 points, and the middle school or above group ≤24 points. Below the threshold is cognitive impairment, above is normal.
MMSE | At the 6 month
  The investigators assessed orientation (10 points), immediate recall (3 points), attention and computation (5 points), delayed recall (3 points), language function (8 points) (naming, retelling, reading, writing, understanding), and visuospatial perception (1 point). The total score is 30 points, and the demarcation between normal and abnormal is related to education level: the uneducated ≤17 points, the primary school group ≤6 years of education ≤20 points, and the middle school or above group ≤24 points. Below the threshold is cognitive impairment, above is normal.
MMSE | At the 12 month
  The investigators assessed orientation (10 points), immediate recall (3 points), attention and computation (5 points), delayed recall (3 points), language function (8 points) (naming, retelling, reading, writing, understanding), and visuospatial perception (1 point). The total score is 30 points, and the demarcation between normal and abnormal is related to education level: the uneducated ≤17 points, the primary school group ≤6 years of education ≤20 points, and the middle school or above group ≤24 points. Below the threshold is cognitive impairment, above is normal.
Digital Sign Conversion Test | Baseline
  The subjects are required to be familiar with nine different symbols representing the nine numbers from 1 to 9, and then they are asked to fill in the corresponding symbols according to the given numbers as much as possible in the 90s. The exact number recorded is the score.
Digital Sign Conversion Test | At the 6 month
  The subjects are required to be familiar with nine different symbols representing the nine numbers from 1 to 9, and then they are asked to fill in the corresponding symbols according to the given numbers as much as possible in the 90s. The exact number recorded is the score.
Digital Sign Conversion Test | At the 12 month
  The subjects are required to be familiar with nine different symbols representing the nine numbers from 1 to 9, and then they are asked to fill in the corresponding symbols according to the given numbers as much as possible in the 90s. The exact number recorded is the score.
Reverse digit recitation | Baseline
  A series of 1-9 digits are orally reported to the subject at the rate of one per second. The subject needs to quickly retell the whole string of digits in reverse order after the subject stops counting. The shortest sequence consists of three digits, and there are two sequences of each length. If the subject answers at least one sequence correctly, the sequence length is increased by one, otherwise the test ends. If both sequences of the maximum length that the subject can answer correctly are answered correctly, the length is recorded as the number memory span of the subject; if only one sequence is answered correctly, the length minus 0.5 is recorded as the number memory span of the subject.
Reverse digit recitation | At the 6 month
  A series of 1-9 digits are orally reported to the subject at the rate of one per second. The subject needs to quickly retell the whole string of digits in reverse order after the subject stops counting. The shortest sequence consists of three digits, and there are two sequences of each length. If the subject answers at least one sequence correctly, the sequence length is increased by one, otherwise the test ends. If both sequences of the maximum length that the subject can answer correctly are answered correctly, the length is recorded as the number memory span of the subject; if only one sequence is answered correctly, the length minus 0.5 is recorded as the number memory span of the subject.
Reverse digit recitation | At the 12 month
  A series of 1-9 digits are orally reported to the subject at the rate of one per second. The subject needs to quickly retell the whole string of digits in reverse order after the subject stops counting. The shortest sequence consists of three digits, and there are two sequences of each length. If the subject answers at least one sequence correctly, the sequence length is increased by one, otherwise the test ends. If both sequences of the maximum length that the subject can answer correctly are answered correctly, the length is recorded as the number memory span of the subject; if only one sequence is answered correctly, the length minus 0.5 is recorded as the number memory span of the subject.
N-back task | Baseline
  Subjects compare the previous stimulus with the NTH stimulus. When n=1, subjects are asked to compare the current stimulus with the previous stimulus adjacent to it. When n=2, the current stimulus is compared with the stimulus in the other position. When n=3, the investigators want to compare the current stimulus with the stimulus two positions away from it. Finally, the response time and discrimination of subjects under different memory loads were counted.
N-back task | At the 6 month
  Subjects compare the previous stimulus with the NTH stimulus. When n=1, subjects are asked to compare the current stimulus with the previous stimulus adjacent to it. When n=2, the current stimulus is compared with the stimulus in the other position. When n=3, the investigators want to compare the current stimulus with the stimulus two positions away from it. Finally, the response time and discrimination of subjects under different memory loads were counted.
N-back task | At the 12 month
  Subjects compare the previous stimulus with the NTH stimulus. When n=1, subjects are asked to compare the current stimulus with the previous stimulus adjacent to it. When n=2, the current stimulus is compared with the stimulus in the other position. When n=3, the investigators want to compare the current stimulus with the stimulus two positions away from it. Finally, the response time and discrimination of subjects under different memory loads were counted.
Structural MRI | Baseline
  Sagittal scan, TR = 8.16ms, TE = 3.18ms, FA= 8O, data size: 256×256×1176, resolution 1×1×1mm3.
Structural MRI | At the 6 month
  Sagittal scan, TR = 8.16ms, TE = 3.18ms, FA= 8O, data size: 256×256×1176, resolution 1×1×1mm3.
Structural MRI | At the 12 month
  Sagittal scan, TR = 8.16ms, TE = 3.18ms, FA= 8O, data size: 256×256×1176, resolution 1×1×1mm3.
Resting state fMRI | Baseline
  Axial scanning, TR = 2000ms, TE = 30ms, 43 layers, resolution 3.42×3.42, rotation Angle (FA) = 90o, FOV = 240mm, layer thickness = 3.2mm, layer spacing =0mm.
Resting state fMRI | At the 6 month
  Axial scanning, TR = 2000ms, TE = 30ms, 43 layers, resolution 3.42×3.42, rotation Angle (FA) = 90o, FOV = 240mm, layer thickness = 3.2mm, layer spacing =0mm.
Resting state fMRI | At the 12 month
  Axial scanning, TR = 2000ms, TE = 30ms, 43 layers, resolution 3.42×3.42, rotation Angle (FA) = 90o, FOV = 240mm, layer thickness = 3.2mm, layer spacing =0mm.
Task state fMRI | Baseline
  Axial scanning, TR = 2000ms, TE = 30ms, 43 layers, resolution 3.42×3.42, rotation Angle (FA) = 90o, FOV = 240mm, layer thickness = 3.2mm, layer spacing =0mm.
Task state fMRI | At the 6 month
  Axial scanning, TR = 2000ms, TE = 30ms, 43 layers, resolution 3.42×3.42, rotation Angle (FA) = 90o, FOV = 240mm, layer thickness = 3.2mm, layer spacing =0mm.
Task state fMRI | At the 12 month
  Axial scanning, TR = 2000ms, TE = 30ms, 43 layers, resolution 3.42×3.42, rotation Angle (FA) = 90o, FOV = 240mm, layer thickness = 3.2mm, layer spacing =0mm.
Arterial spin labeling | Baseline
  3D pCASL sequence; Thick = 3 mm; 45 layer; TR=4781ms; TE = 11.12 ms; TI=1525ms; The size of axial position matrix is 128×128. Axial image resolution 1.72×1.72 mm2; FA =111 o; Marking time 1500 ms; The total scanning time is 6 minutes and 48 seconds.
Arterial spin labeling | At the 6 month
  3D pCASL sequence; Thick = 3 mm; 45 layer; TR=4781ms; TE = 11.12 ms; TI=1525ms; The size of axial position matrix is 128×128. Axial image resolution 1.72×1.72 mm2; FA =111 o; Marking time 1500 ms; The total scanning time is 6 minutes and 48 seconds.
Arterial spin labeling | At the 12 month
  3D pCASL sequence; Thick = 3 mm; 45 layer; TR=4781ms; TE = 11.12 ms; TI=1525ms; The size of axial position matrix is 128×128. Axial image resolution 1.72×1.72 mm2; FA =111 o; Marking time 1500 ms; The total scanning time is 6 minutes and 48 seconds.
Incidence of cardiac events | At the 6 month
  Long-term cardiac events in this study included stroke, heart failure, acute myocardial infarction and sudden cardiac death.
Incidence of cardiac events | At the 12 month
  Long-term cardiac events in this study included stroke, heart failure, acute myocardial infarction and sudden cardiac death.

CONTACTS AND LOCATIONS:
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China